CLINICAL TRIAL: NCT05044793
Title: A Multicenter Clinical Study To Assess The Long-Term Safety And Effectiveness Of The OMNI® Surgical System In Combination With Cataract Surgery In Eyes With Open Angle Glaucoma (GEMINI 2.0)
Brief Title: A Clinical Study To Assess The Safety And Effectiveness Of The OMNI® Surgical System
Status: Completed | Type: Observational
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 07408
Record Dates: First submitted 2021-09-09; First posted 2021-09-16 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Cohort A: Subjects who had a surgical washout of ocular hypotensive medications with post-washout DIOP of 21-36mmHg and were treated with OMNI Surgical System for OAG in combination with cataract extraction at least 700 days prior to study enrollment.
  Interventions: Device: OMNI® Surgical System
- Cohort B: Subjects without a surgical washout of ocular hypotensive medications with pre-surgical medicated IOP≥18 mmHg and on 1 to 5hypotensive medications and were treated with OMNI Surgical System for OAG in combination with cataract extraction at least 700 days prior to study enrollment.
  Interventions: Device: OMNI® Surgical System

INTERVENTIONS:
Device: OMNI® Surgical System — The OMNI® Surgical System is indicated for canaloplasty (microcatheterization and transluminal viscodilation of Schlemm's canal) followed by trabeculotomy (cutting of trabecular meshwork) to reduce intraocular pressure in adult patients with primary open-angle glaucoma.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and effectiveness of the OMNI® Surgical System in subjects who were treated under protocol #06213

ELIGIBILITY:
Inclusion Criteria:

• Participated in, received treatment, and completed Protocol #06213

Exclusion Criteria:

* Systemic disease that, in the opinion of the Investigator, would put the subject's health at risk and/or prevent completion of required study visits
* Ocular pathology which, in the Investigator's judgment, would either place the subject at increased risk of complications, contraindicate washout, place the subject at risk of significant vision loss during the study period (e.g., wet age macular degeneration (AMD), corneal edema, Fuch's dystrophy, active intraocular infection or inflammation within 30 days prior to Screening Visit, etc.), or interfere with compliance to elements of the study protocol (e.g., returning to Investigator's office for follow-up visits)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who received treatment and completed Protocol #06213
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Grene Vision Group, Wichita, Kansas
  - Oklahoma Eye Surgeons, Oklahoma City, Oklahoma
  - Northern Ophthalmics, Jenkintown, Pennsylvania
  - El Paso Eye Surgeons, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Subjects who had a pre-surgical washout of ocular hypotensive medications with post-washout DIOP of 21-36mmHg and were treated with OMNI Surgical System for OAG in combination with cataract extraction at least 700 days prior to study enrollment.
- Cohort B: Subjects without a pre-surgical washout of ocular hypotensive medications with pre-surgical medicated IOP≥18 mmHg and on 1 to 5 hypotensive medications and were treated with OMNI Surgical System for OAG in combination with cataract extraction at least 700 days prior to study enrollment.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 66 | 4
Completed | 66 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) analysis population included all subjects who were enrolled and treated, regardless of whether or not they had a protocol deviation
Groups:
- Cohort A: Pre-operative washout of ocular hypotensive medications with post-washout DIOP of 21-36mmHg
- Cohort B: No pre-operative washout of ocular hypotensive medications with pre-operative medicated IOP ≥18 mmHg and on 1 to 5 hypotensive medications
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 66 | 4 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 1 | 14
  >=65 years | 53 | 3 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at consent
  years | 71.6 (7.5) | 68.0 (14.1) | 71.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 2 | 38
  Male | 30 | 2 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 1 | 23
  Not Hispanic or Latino | 44 | 3 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 59 | 4 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 4 | 70

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: Rate of occurrence of sight-threatening adverse events
Time Frame: 12 months
Population: ITT/Safety population
Measure: Mean (Standard Deviation); unit: adverse event
Groups:
- Cohort A: Pre-operative washout of ocular hypotensive medications.
- Cohort B: No pre-operative washout of ocular hypotensive medications.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 66 | 4
adverse event | 0 (0) | 0 (0)

2. Other Pre Specified Outcome: Change in Intraocular Pressure (IOP)
Description: Mean change in IOP
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Cohort A: Reduction in mean unmedicated diurnal IOP (DIOP) from the preoperative unmedicated DIOP
- Cohort B: Reduction in mean medicated IOP from pre-operative medicated IOP
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 66 | 4
mmHg | -6.89 (3.42) | -11.00 (16.45)

3. Other Pre Specified Outcome: Change in Hypotensive Medications
Description: Reduction in number of hypotensive medications from baseline to 36 months
Time Frame: 12 months
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: number of medications
Groups:
- Cohort A: Reduction in mean number of IOP lowering medications from pre-washout (pre-surgical) baseline at 36 months
- Cohort B: Reduction in mean number of IOP lowering medications from pre-surgical baseline at 36 months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 66 | 4
number of medications | -1.2 (0.87) | -1.0 (1.00)

4. Other Pre Specified Outcome: Number of Participants With ≥20% Reduction in IOP From Baseline to 36 Months
Description: For subjects in cohort A : ≥20% reduction in unmedicated diurnal IOP from baseline to 36 months For subjects in cohort B: ≥20% reduction in mean medicated IOP from baseline to 36 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: ≥20% reduction in unmedicated diurnal IOP from baseline to 36 months
- Cohort B: ≥20% reduction in mean medicated IOP from baseline to 36 months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 66 | 4
Participants | 45 | 1

5. Other Pre Specified Outcome: Number of Participants With Intraocular Pressure (IOP) Between 6 and 18mmHg Inclusive.
Description: For cohort A: unmedicated diurnal IOP between 6 and 18 mmHg inclusive For cohort B: medicated IOP between 6 and 18 mmHg inclusive
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Unmedicated diurnal IOP between 6 and 18 mmHg inclusive
- Cohort B: Medicated IOP between 6 and 18 mmHg inclusive
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 66 | 4
Participants | 41 | 2

ADVERSE EVENTS:
Time Frame: 36 months
Description: Adverse events were collected from the time of the study procedure (retrospective data) through the 36-month visit.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/4
Other Adverse Events (participants affected / at risk) | 27/66 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=66) | Cohort B (N=4)
Adverse events (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fell and cracked hip. Surgery required.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=66) | Cohort B (N=4)
Ocular adverse events (Eye disorders) | 27 (35) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution or PI will submit a copy of any proposed publication/disclosure to Sponsor, at least sixty (60) days prior to submission. Sponsor may request changes or other measures to ensure the information is fairly stated. At Sponsor's request the Institution and/or the PI shall not publish/disclose information related to the Study. If Sponsor indicates that such publication or disclosure contains Confidential Information, the Institution and PI agree to remove such Confidential Information

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT05044793/Prot_SAP_000.pdf